CLINICAL TRIAL: NCT03698370
Title: 68Ga-NeoBOMB1 and 68Ga-PSMA R2 PET/MRI in the Evaluation of Patients With Biochemical Recurrence of Prostate Cancer
Brief Title: Gallium Ga 68 DOTA-NeoBOMB1 and Gallium Ga 68 PSMA-R2 PET/MRI in Diagnosing Participants With Recurrent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andrei Iagaru (Other)
Responsible Party: Sponsor-Investigator, Andrei Iagaru, Professor of Radiology (Nuclear Medicine), Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-46258; NCI-2018-01799 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB-46258 (Other: Stanford IRB); PROS0089 (Other: OnCore ID)
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Prostate Adenocarcinoma; PSA Progression; Recurrent Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm I (Ga68-NeoBOMB1 and Ga68 PSMA-R2 (Experimental): Participants receive gallium Ga 68 DOTA-NeoBOMB1 IV and 45 minutes later, undergo PET/MRI. Within 2 weeks, participants receive gallium Ga 68 PSMA-R2 IV then undergo PET/MRI 45-60 minutes later.
  Interventions: Drug: Gallium Ga 68 DOTA-NeoBOMB1; Device: Gallium Ga 68 PSMA-R2
- Arm II (Ga68 PSMA-R2 and Ga 68-NeoBOMB1) (Experimental): Participants receive gallium Ga 68 PSMA-R2 IV and 45-60 minutes later undergo PET/MRI. Within 2 weeks, participants receive gallium Ga 68 DOTA-NeoBOMB1 IV then undergo PET/MRI 45 minutes later.
  Interventions: Drug: Gallium Ga 68 DOTA-NeoBOMB1; Device: Gallium Ga 68 PSMA-R2

INTERVENTIONS:
Drug: Gallium Ga 68 DOTA-NeoBOMB1 — Administered intravenously (IV)
  Other Names: Ga68-NeoBOMB1
Device: Gallium Ga 68 PSMA-R2 — Administered intravenously (IV)
  Other Names: Ga68 PSMA-R2

SUMMARY:
This phase II trial studies how well gallium Ga 68 DOTA-NeoBOMB1 and gallium Ga 68 PSMA-R2 positron emission tomography (PET)/magnetic resonance imaging (MRI) work in diagnosing participants with prostate cancer that has come back. Diagnostic procedures, such as gallium Ga 68 DOTA-NeoBOMB1 and gallium Ga 68 PSMA-R2 PET/MRI, may help find and diagnose prostate cancer and find out how far the disease has spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate gallium Ga 68 DOTA-NeoBOMB1 (68Ga-NeoBOMB1) and gallium Ga 68 PSMA-R2 (68Ga-PSMA R2) PET/MRI for detection of recurrent prostate cancer after initial therapy in patients meeting the criterion of biochemical recurrence.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive gallium Ga 68 DOTA-NeoBOMB1 intravenously (IV) and 45 minutes later, undergo PET/MRI. Within 2 weeks, participants receive gallium Ga 68 PSMA-R2 IV then undergo PET/MRI 45-60 minutes later.

ARM II: Participants receive gallium Ga 68 PSMA-R2 IV and 45-60 minutes later undergo PET/MRI. Within 2 weeks, participants receive gallium Ga 68 DOTA-NeoBOMB1 IV then undergo PET/MRI 45 minutes later.

After completion of study, participants are followed up at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven prostate adenocarcinoma.
* Rising prostate-specific antigen (PSA) after definitive therapy with prostatectomy or radiation therapy (external beam or brachytherapy).

  a. Post radical prostatectomy (RP) - American Urological Association (AUA) recommendation.

  (i) PSA greater than 0.2 ng/mL measured after at least 6 weeks from radical prostatectomy.

(ii) Confirmatory persistent PSA greater than 0.2 ng/mL (total of two PSA measurements greater than 0.2 ng/mL).

b. Post-radiation therapy ? American Society for Therapeutic Radiology and Oncology (ASTRO)-Phoenix consensus definition.

(i) A rise of PSA measurement of 2 or more ng/mL over the nadir.

* Able to provide written consent.
* Karnofsky performance status of >= 50 (or Eastern Cooperative Oncology Group [ECOG]/World Health Organization [WHO] equivalent).

Exclusion Criteria:

* Inability to lie still for the entire imaging time.
* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.).
* Any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance.
* Known allergy, hypersensitivity, or intolerance to the investigational product or its excipients.
* Metallic implants (contraindicated for magnetic resonance imaging [MRI]).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, Principal Investigator — Stanford Cancer Institute Palo Alto
Locations (1):
- Stanford Cancer Institute Palo Alto, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ga68-NeoBOMB1 Then Ga68 PSMA-R2: Participants receive gallium Ga 68 DOTA-NeoBOMB1 IV and 45 minutes later, undergo PET/MRI. Within 2 weeks, participants receive gallium Ga 68 PSMA-R2 IV then undergo PET/MRI 45-60 minutes later.
- Ga68 PSMA-R2 Then Ga 68-NeoBOMB1): Participants receive gallium Ga 68 PSMA-R2 IV and 45-60 minutes later undergo PET/MRI. Within 2 weeks, participants receive gallium Ga 68 DOTA-NeoBOMB1 IV then undergo PET/MRI 45 minutes later.
Period: First Scan
Arm/Group | Ga68-NeoBOMB1 Then Ga68 PSMA-R2 | Ga68 PSMA-R2 Then Ga 68-NeoBOMB1)
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0
Period: Second Scan
Arm/Group | Ga68-NeoBOMB1 Then Ga68 PSMA-R2 | Ga68 PSMA-R2 Then Ga 68-NeoBOMB1)
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ga68-NeoBOMB1 Then Ga68 PSMA-R2 | Ga68 PSMA-R2 Then Ga 68-NeoBOMB1) | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (8.1) | 67.9 (9.4) | 67.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 11 | 14 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 11 | 12 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Lesions Detected by Investigational Imaging Agent
Description: The number of lesions detected on Ga- NeoBOMB1 positron emission tomography (PET)/magnetic resonance imaging (MRI), Ga PSMA R2 PET/MRI, and conventional MR will be compared.
Time Frame: Up to approximately 2 hours to complete each scan
Measure: Number; unit: lesions
Groups:
- Ga68-NeoBOMB1: Participants receive gallium Ga 68 DOTA-NeoBOMB1.
- Ga68 PSMA-R2: Participants receive gallium Ga 68 PSMA-R2.
Arm/Group | Ga68-NeoBOMB1 | Ga68 PSMA-R2
Number analyzed (Participants) | 27 | 27
lesions | 31 | 20

2. Secondary Outcome: Number of Detected Lesions Confirmed to be Malignant for Each Imaging Method
Description: The predictive value of Ga- NeoBOMB1 PET/MRI and Ga PSMA R2 PET/MRI imaging will be evaluated based on biopsy and/or imaging results at the end of the 12 month standard clinical follow-up period, by comparing the investigational scans against scans the patient received as standard of care.
Time Frame: At 1 year post-scan follow-up
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Ga68-NeoBOMB1 | Ga68 PSMA-R2
Number analyzed (Participants) | 27 | 27
Number analyzed (lesions) | 31 | 20
lesions | 18 | 15

ADVERSE EVENTS:
Time Frame: 2 weeks, plus safety follow up at to 72 hours after the final scan
Groups:
- Ga68-NeoBOMB1: 68Ga-NeoBOMB1 PET/MRI for detection of recurrent prostate cancer.
- Ga68 PSMA-R2: Ga68 PSMA-R2 PET/MRI for detection of recurrent prostate cancer.
Arm/Group | Ga68-NeoBOMB1 | Ga68 PSMA-R2
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT03698370/Prot_SAP_000.pdf